CLINICAL TRIAL: NCT06761222
Title: The Impact of Ultrasound Use in Central Block Applications in Obstetric Anesthesia
Brief Title: Impact of Ultrasound in Obstetric Anesthesia Central Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sukran Ozbebek, Anesthesiologist, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-6.2/4
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia
Keywords: Regional Anesthesia; Central Block; Obstetrics; Ultrasound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- obstetric patient (Experimental): Regional block procedures were performed on all patients included in the study in a sitting position, using the most appropriate interspinous space among L3-L4-L5-S1. Ultrasonography was conducted using a convex probe in the paramedian and transverse planes, and the images were recorded. Regional (spinal and/or epidural) anesthesia was provided by entering the lumbar space identified with ultrasonography.
  Interventions: Other: The use of ultrasound in central blocks

INTERVENTIONS:
Other: The use of ultrasound in central blocks — Ultrasonography was conducted using a convex probe in the paramedian and transverse planes.

SUMMARY:
This study aimed to evaluate the use of ultrasound in obstetric anesthesia, specifically for measuring epidural and intrathecal distances in pregnant women undergoing cesarean section. The relationship between skin-subdural distance (Ultrasound depth) and needle depth was assessed, and the accuracy of ultrasound in determining needle entry site, needle distance, trial attempts, and block success was examined. Additionally, complications such as paresthesia, lower back pain, and postoperative headache were queried and recorded.

DETAILED DESCRIPTION:
Obstetric anesthesia generally posed low risks; however, the difficulty of the procedure and the potential complications increased due to the anatomical and physiological changes associated with pregnancy.

The aim of study was to measure epidural and intrathecal distances in pregnant women undergoing cesarean sections and to evaluate the relationship between the skin-subdural distance (Ultrasound depth) and needle depth. The investigator assessed the accuracy of Ultrasound in determining the needle entry site, needle distance (measured at the site where cerebrospinal fluid flow occurred or where there was a loss of resistance in the epidural space), trial numbers, and block success. Additionally, occurrences of paresthesia and lower back pain during the procedure, as well as postoperative headaches following dural puncture, were queried and recorded.

After obtaining approval from the Ege University Faculty of Medicine Ethical Committee, the study was prospectively conducted in the operating room of the Department of Obstetrics and Gynecology at Ege University Hospital. One hundred pregnant women classified as ASA I-II, between 37-42 gestational weeks, undergoing elective cesarean sections with neuraxial blocks (spinal and/or epidural), were included after obtaining their consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as ASA I-II
* Patients at 37-42 gestational weeks
* Patients scheduled for elective cesarean section under neuraxial block (spinal and/or epidural)

Exclusion Criteria:

* Patients who did not consent to spinal anesthesia
* Patients with contraindications for regional anesthesia (coagulopathy, local or systemic infection)
* Emergency patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Investigating The Skin-to-subdural/epidural Distance and Needle Depth in Central Block applications | Preoperative
  The Use of Ultrasonography in Central Block Applications in Obstetric Patients

CONTACTS AND LOCATIONS:
Overall Officials: Şükran ÖZBEBEK, MD, Study Director — Ege Univesity
Locations (1):
- Şükran Özbebek, Izmir, Turkey (Türkiye)